CLINICAL TRIAL: NCT06890429
Title: Randomized, Double-blind, Placebo-controlled Phase 2 Trial of RSV/Flu-01E Vaccine for the Prevention of Respiratory Syncytial Virus Infection in Volunteers Over 60 Years
Brief Title: Phase 2 Study of the RSV/Flu-01E Vaccine Against Respiratory Syncytial Virus Infection in Older Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Research Institute of Influenza, Russia (Other)
Collaborators: Pavlov First Saint Petersburg State Medical University (Other); St. Petersburg City Polyclinic No. 34 (Unknown)
Responsible Party: Principal Investigator, Tatyana Zubkova, Head of the clinical department, Research Institute of Influenza, Russia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RSV-II-06/2023
Record Dates: First submitted 2025-03-17; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2023-11

CONDITIONS: Respiratory Synctial Virus Infections
Keywords: Respiratory syncytial virus infection; Mucosal Vaccine; Influenza Vector; Intranasal Immunization
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RSV/Flu-01E (Experimental): Single dose of RSV/Flu-01E vector vaccine
  Interventions: Biological: RSV/Flu-01E
- Placebo (Placebo Comparator): Single dose of Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: RSV/Flu-01E — Participants will receive single intranasal injection of RSV/Flu-01E vaccine in 0.5 ml, containing 8.4 lg EID50 of A/H1N1pdm09 recombinant attenuated influenza vector with modified NS gene, encoding for the F antigen of respiratory syncytial virus
  Arms: RSV/Flu-01E
Other: Placebo — Participants will receive single intranasal injection of physiological buffer solution in 0.5 ml
  Arms: Placebo

SUMMARY:
The aim of the study is to investigate immunogenicity and safety of the RSV/Flu-01E intranasal vaccine for the prevention of respiratory syncytial virus infection in volunteers over 60 years

DETAILED DESCRIPTION:
Study includes 120 participants over 60 years randomized at 3:1 ratio, to receive single intranasal dose of RSV/Flu-01E vaccine or placebo, correspondingly. Duration of the study for each participant is about 4 months (118±3 days)

ELIGIBILITY:
Inclusion Criteria:

1. Availability of signed informed consent
2. Adult men and women over the age of 60.
3. The diagnosis is "healthy", verified according to standard clinical, laboratory and instrumental methods of examination or the presence of a chronic disease, if the researcher considers it to be compensated.
4. BMI from 18 to 30 kg/m2.
5. The ability and willingness to make entries in the diary of self-observation, as well as to carry out all the visits foreseen in the study for control medical observation
6. Negative test for alcohol in exhaled air
7. Values of the complete blood count and biochemical blood analysis (during the screening) within 0.9*reference range lower limit and 1,1 * reference range upper limit
8. Negative tests for HIV, hepatitis B, hepatitis C, and syphilis

Exclusion Criteria:

1. Participation in another clinical study within three months prior to the start of the current study; planning to participate in another study during the current study period
2. Contact with COVID-19 patients within 14 days prior to the start of the clinical study
3. Positive rapid test result for SARS-CoV-2 antigen
4. Immunization with any other non-study vaccine product within three weeks prior to enrollment in the current study, or refusal to postpone such until the end of the three-week period after completion of the current study
5. Regular use of nasal irrigation therapy during the last six months prior to enrollment in the current study or episodic use of the above method of treatment in the two weeks prior to the screening
6. History of frequent nosebleeds (>5) during the year prior to the current study
7. Features of the nasal anatomy that may complicate intranasal administration of the study drug
8. Surgical interventions or traumatic injuries in the sinus area, paranasal sinuses, or traumatic injuries of the nose within a month before screening
9. Symptoms of acute respiratory disease, including fever, or other acute illness at the time of screening or within two weeks prior to screening
10. Treatment with immunoglobulins or other blood derived medications in the three months prior to screening or planning such treatment during the period of participation in the current study
11. Donation of blood/plasma (450 ml or more) less than 2 months prior to screening.
12. The presence or suspicion of the presence of various immunosuppressive or immunodeficiency conditions or continuous use (the drug was prescribed for more than 14 days without a break) of immunosuppressive drugs, immunomodulators for 6 months before the screening.
13. History of bronchial asthma
14. Hypersensitivity and the presence of severe allergic reactions, including Quincke's edema, anaphylactic shock after the previous administration of any vaccine
15. History of wheezing after previous immunization with live influenza vaccine
16. Other adverse events after immunization (fever above 40°C, syncope, non-febrile convulsions, anaphylaxis) when there is a minimal likelihood that they are associated with a previous administration of any vaccine
17. Suspicion of hypersensitivity to any component of the study vaccine, including egg protein
18. Acute or chronic clinically significant lung, cardiovascular, hepatic, endocrine, neurological, or psychiatric disorders, or impaired renal function identified by history, physical examination, or clinical laboratory findings that, in the opinion of the investigator, may influence the outcome of the study
19. History of oncological diseases
20. History of thrombocytopenic purpura or bleeding disorders
21. History of convulsions
22. Tuberculosis or residual changes after tuberculosis according to the anamnesis and / or available medical documentation
23. Chronic alcohol dependence or chronic use of illicit drugs, drug abuse
24. Claustrophobia and social phobia according to history and / or available medical records
25. Inability to read Russian; inability or unwillingness to understand the essence of the study
26. Military personnel serving in the military or law enforcement officers.
27. Special diet (eg, vegetarian, vegan, salt-restricted) or lifestyle (night work, extreme physical activity)
28. Any condition that, in the opinion of the investigator, may increase the risk to the health of a volunteer participating in the study or affect the results of the study

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-12-07 (Actual); Primary Completion 2024-01-08 (Actual); Study Completion 2024-04-08 (Actual)

PRIMARY OUTCOMES:
Level of RSV F antigen-specific cytokine producing CD4+ and CD8+ T-cells | Days 1, 7, 28
  Change from baseline in the level of cytokine producing CD4+ and CD8+ T-cells upon in vitro stimulation of PBMC with RSV F-peptide epitopes measured by FACS/ELISPOT
Level of the RSV F antigen-specific Th1/Th2 cytokine release in whole blood assay | Days 1, 7, 28
  Change from the baseline of the cytokine concentration in whole-blood cytokine release assay upon in vitro stimulation with RSV F-peptide epitopes measured in ELISA

SECONDARY OUTCOMES:
Number of participants with local and systemic adverse events (AEs) and serious adverse events (SAEs) | Throughout the study, average 4 months
  Adverse events (AEs) and serious AEs (SAEs), both vaccine related, and non-vaccine related; AEs/SAEs of particular importance:
  * Immediate AEs (allergic reactions) occurring within two hours of vaccination.
  * Post-vaccination reactions (anticipated clinical manifestations of a local and systemic nature), usually due to intranasal vaccination between two hours and the next 7 days after vaccination
Concentration of cytokines in nasal secrets after vaccination | Days 1, 2, 3
  Change from baseline in the concentration of cytokines in nasal secrets measured in ELISA
Level of RSV F antigen-specific IgG antibody in serum | Days 1, 28, 118±3
  Change from the baseline in the level of RSV F antigen-specific serum IgG antibodies measured in ELISA
Influenza specific systemic antibody immune response | Days 1, 28, 118±3
  Change from the baseline in the titer of influenza specific antibodies in serum measured in hemagglutination inhibition/microneutralization assay
Level of mucosal IgA antibody in nasal secret | Days 1, 28
  Change from the baseline in the level of IgA antibody measured in ELISA in nasal secret
Level of influenza specific cytokine release in whole blood assay | Days 1, 7, 28
  Change from the baseline of the cytokine concentration in whole-blood cytokine release assay upon in vitro stimulation with influenza A/H1N1pdm antigen measured in ELISA
Level of B-cell populations | Days 1, 7, 28
  Change from the baseline in the relative amount of B-cell populations in PBMC measured by FACS

CONTACTS AND LOCATIONS:
Overall Officials: Marina Stukova, Dr, Study Director — Smorodintsev Research Institute of Influenza
Locations (3):
- Russia (3):
  - Pavlov First Saint Petersburg State Medical University, Saint Petersburg
  - Smorodintsev Research Institute of Influenza, Saint Petersburg
  - St. Petersburg City Polyclinic No. 34, Saint Petersburg

IPD SHARING:
Plan to Share IPD: Yes
Only IPD used in the results publication will be available
Access Criteria: IPD will be available upon reasonable request to Study Director. Once the request is approved, the data can be transferred via a secure online platform